CLINICAL TRIAL: NCT06327256
Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Oral Doses of BI 3000202 in Healthy Male and Female Subjects (Double-blind, Randomised, Placebo-controlled, Parallel Group Design) and Evaluation of Midazolam Interaction in Healthy Male and Female Subjects (Nested, Open, Fixed-sequence, Intra-individual Comparison)
Brief Title: A Study in Healthy People to Test How Well Different Doses of BI 3000202 Are Tolerated and How They Affect the Way the Body Handles Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 1509-0002; 2023-509293-29-00 (Registry Identifier: CTIS); U1111-1299-6907 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: The multiple rising dose part of the trial will be conducted in a parallel group assignment. The effect of midazolam interaction will be assessed sequentially.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The multiple rising dose part of the trial will be blinded to the participants and investigators . The effect of midazolam will be assessed open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose group 1 (Experimental): Group receiving placebo or dose 1 of BI 3000202
  Interventions: Drug: BI 3000202; Drug: Placebo
- Dose group 2 (Experimental): Group receiving placebo or dose 2 of BI 3000202
  Interventions: Drug: BI 3000202; Drug: Placebo
- Dose group 3 (Experimental): Group receiving midazolam, midazolam and dose 3 of BI 3000202 or midazolam and placebo, and only BI 3000202 or only placebo
  Interventions: Drug: BI 3000202; Drug: Placebo; Drug: Midazolam
- Dose group 4 (Experimental): Group receiving midazolam, midazolam and dose 4 of BI 3000202 or midazolam and placebo, and only BI 3000202 or only placebo
  Interventions: Drug: BI 3000202; Drug: Placebo; Drug: Midazolam

INTERVENTIONS:
Drug: BI 3000202 — BI 3000202
Drug: Placebo — Placebo-matching BI 3000202
Drug: Midazolam — Midazolam
  Arms: Dose group 3; Dose group 4

SUMMARY:
The aim of this trial is to investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) following multiple rising doses of BI 3000202 and to investigate the effect of BI 3000202 on the metabolism of midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female of non-childbearing potential subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m^2 (inclusive)
* Signed and dated written informed consent in accordance with International Conference of Harmonization-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with drug-related adverse events | Up to day 20

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 3000202 in plasma over the dosing interval 0 to 12 hours (AUC0-12) | Up to 12 hours
Maximum measured concentration BI 3000202 in plasma (Cmax) | Up to 24 hours
Area under the concentration-time curve of BI 3000202 in plasma over a uniform dosing interval τ (AUCτ,ss) at steady state | Up to day 20
Maximum measured concentration of BI 3000202 in plasma (Cmax,ss) at steady state | Up to day 20
Time from dosing to the maximum measured concentration of BI 3000202 in plasma (tmax,ss) at steady state | Up to day 20
Area under the concentration-time curve of midazolam in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) after a single dose | Up to 2 days
Maximum measured concentration of midazolam in plasma (Cmax) after a single dose | Up to 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com